CLINICAL TRIAL: NCT00145847
Title: Naltrexone Treatment of Alcohol Abuse in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Steven Batki, M.D., Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUNY UMU IRB # 4800; 1R01AA013655-01A1 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Mental Disorders; Alcohol Abuse; Alcoholism; Alcohol-related Disorders
Keywords: alcohol; schizophrenia; naltrexone
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Alcoholism; Alcohol-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Active Comparator): Naltrexone 50 mg per day, directly administered as 100 mg on Mondays, 100 mg on Wednesdays and 150 mg on Fridays
  Interventions: Drug: Naltrexone or Placebo
- Lactose pill (Placebo Comparator)
  Interventions: Drug: Naltrexone or Placebo

INTERVENTIONS:
Drug: Naltrexone or Placebo — Naltrexone or Placebo 50 mg per day

SUMMARY:
The primary purpose of this study is to determine whether naltrexone is effective in the treatment of alcohol dependence and abuse in patients with schizophrenia and schizoaffective disorder. Hypotheses are as follows:

hypothesis 1: Naltrexone will be more effective than placebo in reducing alcohol use.

hypothesis 2: Patients responding to naltrexone by reducing alcohol use will also show reductions in severity of psychiatric symptoms and utilization of inpatient and emergency psychiatric services.

hypothesis 3: Severity of psychiatric symptoms and amount of service utilization will correlate positively with alcohol use.

DETAILED DESCRIPTION:
The long-term goal of the proposed project is to improve the treatment of alcohol abuse and dependence in patients with schizophrenia and schizoaffective disorder. Alcohol use disorders are common among patients with severe mental illness. It is estimated that there may be as many as 750,000 individuals in the United States with comorbid schizophrenia and alcohol disorders. Alcohol disorder comorbidity requires treatment because it is associated with adverse consequences such as increased rates of hospitalization. Yet, to date, there are no reports of controlled trials testing the efficacy of pharmacological treatments for alcohol abuse or dependence in this population. Naltrexone pharmacotherapy is an effective treatment for alcohol dependence, but it has not been systematically applied to the care of patients with schizophrenia. The specific aims of this study are: To test the efficacy of naltrexone in reducing alcohol use among individuals with schizophrenia and schizoaffective disorder who also have alcohol abuse or dependence. We will test hypothesis 1: Naltrexone will be more effective than placebo in reducing alcohol use. Our primary outcome measure will be the number of drinking days over the course of the treatment trial. To test naltrexone's efficacy in reducing psychiatric symptom severity and medical utilization by reducing alcohol use. We will test hypothesis 2: Patients responding to naltrexone by reducing alcohol use will also show reductions in severity of psychiatric symptoms and utilization of inpatient and emergency psychiatric services. To determine the relationship between a) changes in alcohol use, and b) psychiatric symptom severity and inpatient and emergency service utilization. We will test hypothesis 3: Severity of psychiatric symptoms and amount of service utilization will correlate positively with alcohol use. The proposed research will study a cohort of 150 subjects in a double-blind, randomized, placebo-controlled trial of naltrexone using three times per week directly observed administration of medication. The study will be 6 months in duration, consisting of a 12-week course of naltrexone or placebo plus 3 monthly follow-up interviews after discontinuation of medication. Voucher incentives contingent on attendance will be provided to all subjects to ensure attendance for medication administration. Weekly motivational enhancement counseling sessions will also be provided to all subjects. Study outcomes will consist of self-report and biological measures of alcohol use as well as measures of psychiatric symptom severity and medical service utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 to 69, with a DSM-IV diagnosis of Schizophrenia or Schizoaffective Disorder;
2. DSM-IV diagnosis of Alcohol Abuse or Alcohol Dependence;
3. Level of Drinking: At least four days of drinking in the 30 days prior to consent;
4. Currently prescribed antipsychotic medication;
5. Currently involved in outpatient psychiatric treatment at one of the study sites (Hutchings Psychiatric Center, St. Joseph's Hospital Health Center, VA Medical Center) or at another location in the community at the time of randomization.

Exclusion Criteria:

1. Inability to give adequate informed consent;
2. Currently taking disulfiram (Antabuse) or naltrexone (ReVia/Depade);
3. Current DSM-IV diagnosis of Opioid Dependence or Opioid Abuse;
4. Currently taking ibuprofen or other potentially hepatotoxic medications in amount and/or frequency judged by the Principal Investigator to pose clinically significant added risk of hepatic injury;
5. Current use of prescribed or non-prescribed opioid analgesics, such as methadone, morphine, codeine, heroin, meperidine, and all other opioids.
6. Female patients of childbearing potential who are sexually active, not sterile, and who deny using a form of birth control;
7. Female patients who are pregnant or nursing;
8. Significant unstable medical problems, including any significant unstable psychiatric disorders. The study physician conducting the medical history and physical exam will exclude such clinically unstable individuals;
9. AST levels greater than 3x upper limit of normal;
10. Subjects who do not attend required screening appointments. Subsequent exclusion from the study for reasons related to non-attendance will be based on the judgment of the principal investigator;
11. In need of acute medical detoxification from alcohol in the judgment of the study physician based on results from the Clinical Institute Withdrawal Assessment of Alcohol Scale Based on DSM-III-R (CIWA-AD) and other information obtained;
12. Scheduled surgery within 3 months of intake;
13. Subjects who have pending legal proceedings whose outcome may lead to incarceration within 3 months of intake.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Measures of Alcohol Use | 12 weeks

SECONDARY OUTCOMES:
Psychiatric Symptom Severity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Batki, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (4):
- United States (4):
  - St. Joseph's Mental Health Services, Syracuse, New York
  - Hutchings Psychiatric Center, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Veterans Administration Healthcare Center, Syracuse, New York

REFERENCES:
- [Background] Batki SL, Dimmock JA, Leontieva L, Bowman ML, Gallinger L, Carey KB, Maisto SA, Canfield KM, McMaster T, Schweizer ML; (abstract) (2005) Recruitment and characteristics of alcohol dependent patients with schizophrenia. Alcoholism Clinical and Experimental Research 29 (5:suppl):78A (abstract 428)
- [Background] Batki SL, Dimmock J, Hameed A, Cornell M, Wade M, Albrecht J, Maisto S, Carey K; (2001) Alcohol use measures in naltrexone treatment of alcohol dependence in schizophrenia: Preliminary analysis. Alcoholism Clinical and Experimental Research, 25 (5:suppl.):93A (abstract 522)
- [Background] Batki SL, Dimmock J, Cornell M, Wade M, Carey K, Maisto S. (2002) Directly observed naltrexone treatment of alcohol dependence in schizophrenia: Preliminary analysis. Alcoholism Clinical and Experimental Research 26 (5:suppl.):83A (abstract 470)
- [Background] Batki SL, Dimmock JA, Wade M, Gately PW, Cornell M, Maisto SA, Carey KB, Ploutz-Snyder R. Monitored naltrexone without counseling for alcohol abuse/dependence in schizophrenia-spectrum disorders. Am J Addict. 2007 Jul-Aug;16(4):253-9. doi: 10.1080/10550490701389732. PMID 17661192
- [Background] Carey KB, Leontieva L, Dimmock J, Maisto SA, Batki SL. Adapting Motivational Interventions for Comorbid Schizophrenia and Alcohol Use Disorders. Clin Psychol (New York). 2007 Mar;14(1):39-57. doi: 10.1111/j.1468-2850.2007.00061.x. PMID 19081784
- [Background] Batki, S. L., Dimmock, J. A., Leontieva, L., Bowman, M. L., Gallinger, L., Schweizer, M. L., Carey, K. B., Maisto, S. A., Canfield, K. M., McMaster, T., Ploutz-Snyder, R. (abstract) (2006). Associations among psychiatric symptoms, alcohol severity, and motivation to change in patients with schizophrenia and alcohol use disorders. American Journal on Addictions 15(4):321-322.
- [Background] Batki, S.L., Dimmock, J.A., Leontieva, L., Bowman, M. L., Gallinger, L., Gately, P. W., Carey, K. B., Maisto, S. A., Canfield, K. M., Ploutz-Snyder, R. (abstract) (2006). Co-occurring substance use among patients with alcohol dependence and schizophrenia. Alcoholism Clinical and Experimental Research 30 (6: suppl.):162A (abstract 621)
- [Background] Carey, K.B., Leontieva, L., Dimmock, J., Bowman, M., Gallinger, L., Gately, P., Maisto, S.A., Ploutz-Snyder, R., Batki, S.L. (abstract) (2006). Psychometrics of a short version of the problems assessment for substance-using psychiatric patients (PASSUP-SV) Alcoholism Clinical and Experimental Research 30(6: suppl.):206A (abstract 799)
- [Background] Leontieva, L., Dimmock, J.A., Gately, P., Gallinger, L., Cavallerano, M., DeRycke, S., McMasters, T., Ploutz-Snyder, R., Strutynski, K., Carey, K.B., Maisto, S.A., & Batki, S.L.(abstract). Voucher-based incentives for adherence to research visits in schizophrenia and alcohol dependence.30th Annual Research Society on Alcoholism Meeting, Chicago, IL, USA, July, 2007
- [Background] Leontieva L, Dimmock JA, Gately PW, Gallinger L, Ploutz-Snyder R, Batki SL. Voucher-based incentives for naltrexone treatment attendance in schizophrenia and alcohol use disorders. Psychiatr Serv. 2008 Mar;59(3):310-4. doi: 10.1176/ps.2008.59.3.310. PMID 18308913
- See also: SUNY Upstate Medical University — http://www.upstate.edu